CLINICAL TRIAL: NCT00307294
Title: Phase II Trial of Thalidomide and Doxil® (Doxorubicin HCL Liposome Injection) in Patients With Androgen Independent Prostate Cancer (AIPC) With a Rising PSA While on Chemotherapy
Brief Title: Thalidomide and Doxil® in Patients With Androgen Independent Prostate Cancer (AIPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-078
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2016-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; Androgen; AIPC; Doxil
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Thalidomide; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- thalidomide and doxil (Experimental): Combination of Thalidomide and Doxil
  Interventions: Drug: Thalidomide; Drug: Doxil

INTERVENTIONS:
Drug: Thalidomide — 100 mg PO q day and escalation will occur bt 50 mg every 4 weeks to a maximum of 200mg
  Other Names: Thalomid
Drug: Doxil — On day 1 of each cycle 40 mg/m2 IV over 1 hr every 28 days
  Other Names: doxorubicin liposome

SUMMARY:
The primary objective of this study is to evaluate PSA response rates of the combination of Doxil and Thalidomide in patients with AIPC who have failed chemotherapy. Secondary objectives include: 1) To evaluate the clinical response rate of this combination on measurable disease 2) To evaluate overall survival for this combination.

DETAILED DESCRIPTION:
This is an open label, Phase II trial of thalidomide and Doxil in patients with androgen independent prostate cancer whom have a rising PSA while on chemotherapy. The primary objective of this study is to evaluate PSA response rates of the combination of Doxil and Thalidomide in patients with AIPC who have failed chemotherapy. Secondary objectives include: 1) To evaluate the clinical response rate of this combination on measurable disease (If measurable soft tissue lesions are present on radiological or clinical exam) ; 2) To evaluate overall survival for this combination. There will be between 18 and 35 subjects at least 18 years of age enrolled on this single site study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Confirmed androgen independent prostate cancer with evidence of rising PSA (two successive increases in PSA, at least 4 weeks apart) while on chemotherapy. If the PSA is less than 5, the increase in PSA must be at least 50%. Must also have castrate testosterone levels (<50 ng/ml)
* Patients could not have received more than 2 previous chemotherapy regimens.
* No anthracyclines within the past 6 months.
* No prior single agent thalidomide in the last 12 months. No prior cytotoxic chemotherapy + thalidomide given in conjunction
* Age > 18 years of age
* Performance status ECOG 0-2
* Peripheral neuropathy must be < grade 1
* Must have adequate hematologic, hepatic and renal function
* Men of reproductive potential must be willing to consent to using effective contraception while on treatment and for at least 4 weeks thereafter
* Patients must have left ventricular ejection fraction of > 50% within 42 days prior to first dose of study drug. The method used at baseline must be used for later monitoring
* Must have been off an anti-androgen for at least 4-6 weeks (Flutamide and Bicalutamide respectively) and documented as having a rising PSA
* Measurable or evaluable disease (PSA elevation will constitute evaluable disease). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques CT scan or as >10 mm with spiral CT scan. See section 6.B for the evaluation of measurable disease
* Life expectancy of greater than 3 months
* Patients must be willing and able to comply with the FDA-mandated S.T.E.P.S.® program
* Ability to understand and sign written informed consent approved by the Institutional Review Board [IRB/Ethics Committee], which will be obtained prior to study entry.

Exclusion Criteria:

* Patients with unstable angina, uncompensated CHF, a history of an MI, PE or DVT within the last 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal S Chatta, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thalidomide and Doxil
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thalidomide and Doxil
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 70 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The number of patients experiencing a response to treatment, per RECIST criteria / total number of patients evaluable for response.
Time Frame: 24 weeks
Population: Patients that received greater than one cycle of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Thalidomide and Doxil
Number analyzed (Participants) | 32
percentage of participants | 9.3 [2 to 25]

2. Secondary Outcome: Best Overall PSA Response
Description: PSA response as stable disease or progressive disease, per Prostate-Specific Antigen Working Group criteria.
Time Frame: 4 weeks
Population: Patients that received greater than one cycle of therapy and met criteria for stable or progressive disease according to Prostate-Specific Antigen Working Group criteria.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Thalidomide and Doxil
Number analyzed (Participants) | 32
percentage of patients
  Stable disease | 48.8 [20 to 60]
  Progressive Disesase | 43.7 [26 to 60]

3. Secondary Outcome: Overall Survival
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide and Doxil
Number analyzed (Participants) | 39
months | 12 [7.9 to 18.9]

4. Secondary Outcome: Time to Progression
Description: Time from start of treatment until the disease progression per RECIST criteria.
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide and Doxil
Number analyzed (Participants) | 39
months | 3.7 [2.2 to 5.5]

ADVERSE EVENTS:
Arm/Group | Thalidomide and Doxil
Serious Adverse Events (participants affected / at risk) | 9/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide and Doxil (N=39)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Edema: limb (General disorders) | 1
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
Pain - Other (General disorders) | 1
Pain, Bone (Musculoskeletal and connective tissue disorders) | 1
Pain, Intestine (Gastrointestinal disorders) | 1
Pain, Pelvis (Gastrointestinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide and Doxil (N=39)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 3
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 18
Leukocytes (total WBC) (Investigations) | 10
Lymphopenia (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7
Platelets (Investigations) | 2
Cardiac Arrhythmia - Other (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Sinus bradycardia (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Supraventricular tachycardia (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 3
Constitutional Symptoms - Other (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 25
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4
Insomnia (Psychiatric disorders) | 1
Rigors/chills (General disorders) | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2
Weight gain (Investigations) | 1
Weight loss (Investigations) | 5
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1
Hot flashes/flushes (Vascular disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 9
Constipation (Gastrointestinal disorders) | 21
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, GU, Urinary NOS (Renal and urinary disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Nose (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 1
Infection with Grade 3 or 4 neutrophils , Lung (pneumonia) (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Dental-tooth (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Oral cavity-gums (gingivitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Sinus (Infections and infestations) | 3
Infection with unknown ANC, Sinus (Infections and infestations) | 1
Edema: limb (General disorders) | 13
Lymphatics - Other (Blood and lymphatic system disorders) | 3
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Alkaline phosphatase (Investigations) | 2
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Extraocular (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 8
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mood alteration, Anxiety (Psychiatric disorders) | 1
Mood alteration, Depression (Psychiatric disorders) | 3
Neurology - Other (Nervous system disorders) | 5
Neuropathy: motor (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 14
Somnolence/depressed level of consciousness (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 4
Ocular/Visual - Other (Eye disorders) | 2
Vision-blurred vision (Eye disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Pain - Other (General disorders) | 4
Pain, Abdomen NOS (Gastrointestinal disorders) | 2
Pain, Back (Musculoskeletal and connective tissue disorders) | 6
Pain, Bone (Musculoskeletal and connective tissue disorders) | 1
Pain, Chest wall (Respiratory, thoracic and mediastinal disorders) | 1
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain, Face (General disorders) | 2
Pain, Head/headache (Nervous system disorders) | 2
Pain, Joint (Musculoskeletal and connective tissue disorders) | 9
Pain, Oral cavity (Gastrointestinal disorders) | 1
Pain, Pelvis (Gastrointestinal disorders) | 1
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Edema, larynx (General disorders) | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 4
Urinary frequency/urgency (Renal and urinary disorders) | 3
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Urine color change (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No